CLINICAL TRIAL: NCT01249833
Title: Randomised, Open-label, Multi-Centre, Phase IV Study Assessing the Effect of Oseltamivir Treatment on Cognitive Function in Subjects With Confirmed Influenza Virus Infection
Brief Title: Effect of Oseltamivir on Cognitive Function in Subjects With Influenza
Acronym: FOCUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trial Management Group Inc. (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAI-001-10
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Influenza
Keywords: Influenza; Cognition; Attention; Simple Reaction Time; Alertness; Calmness; Contentment; Mood
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oseltamivir (Active Comparator): Added to standard of care for influenza
  Interventions: Drug: Oseltamivir
- Standard of care alone (No Intervention): Standard of care for influenza

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir 75mg BID for 5 days
  Other Names: Tamiflu
  Arms: Oseltamivir

SUMMARY:
This study has been designed to determine if subjects treated with oseltamivir in addition to standard of care treatment for influenza demonstrate a greater improvement in attention / working memory / processing speed / mood as compared to subjects receiving standard of care alone. The cognitive tests employed are objective measures developed and administered online by HeadMinder Inc.

DETAILED DESCRIPTION:
Primary Objective:

To determine if subjects treated with oseltamivir in addition to standard of care treatment for influenza demonstrate a greater improvement in attention as compared to subjects receiving standard of care alone.

Secondary Objectives:

To determine if subjects treated with oseltamivir in addition to standard of care treatment for influenza demonstrate a greater improvement in working memory and processing speed as compared to subjects receiving standard of care alone.

Supportive Objectives:

1. To determine if subjects treated with oseltamivir in addition to standard of care treatment for influenza demonstrate a greater improvement in self-rated alertness as compared to subjects receiving standard of care alone.
2. To determine if subjects treated with oseltamivir in addition to standard of care treatment for influenza demonstrate a greater improvement in self-rated calmness and contentment as compared to subjects receiving standard of care alone.
3. To determine if there is a correlation between the rate of improvement in symptom scores and the rate of change in attention and working memory.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, 18 - 65 years of age (inclusive)
2. Indicative symptoms/signs of uncomplicated acute illness due to influenza infection (A or B strains) that started within a maximum of 2 days prior to Visit 1 as per the Tamiflu® Canadian product label. Signs and symptoms may include the following:

   * Fever
   * Respiratory symptoms (cough, coryza, sore throat, rhinitis)
   * Constitutional symptoms (headache, malaise, myalgia, sweats and/or chills, fatigue)
3. Positive rapid antigen test for influenza (A or B strains) at Visit 1
4. Negative urine pregnancy test at Visit 1 for women of childbearing potential; women of childbearing potential who are sexually active must agree to use a suitable form of contraception during the study. Acceptable birth control measures include: hysterectomy, birth control pills, tubal ligation, intrauterine device, hormonal injections and implants, double barrier methods (such as a condom with a diaphragm or a condom with spermicide), and abstinence. Oral contraceptives must be in stable use for 2 or more cycles prior to screening. Intrauterine device (IUD) must be in use at least 30 days prior to study drug administration. Barrier methods must be in use at least 14 days prior to study drug administration.
5. Subjects must:

   * have daily access to a computer at home with: internet access (preferably high-speed for optimal performance but dial-up can be used as well); Microsoft operating system; Internet Explorer browser capability and an e-mail account. A Macintosh (Mac) computer cannot be used.
   * be capable of and willing to complete the required online assessments in English according to the protocol schedule
   * be willing to abstain from the use of an antiviral medication if they are randomised to the standard of care treatment arm
   * have provided written informed consent prior to the initiation of any study procedures

Exclusion Criteria:

1. More than 2 days since the onset of influenza symptoms
2. Subjects who, in the Investigator's judgment, require treatment with an antiviral medication as per the Canadian "Clinical Recommendations for Patients Presenting with Respiratory Symptoms During the 2009 - 2010 Influenza Season" (see Appendix D)
3. Clinical suspicion of infection with a respiratory virus other than influenza
4. Any medical condition that is sufficiently severe or unstable such that the subject is considered to be at imminent risk of requiring hospitalisation
5. History of conditions that may potentially affect cognitive function during the study, such as underlying neurologic conditions, depression or depressive disorders (unless the condition and treatment have been stable for 3 months), seasonal affective disorder (SAD), or any other cognitive impairment or dementia
6. Intermittent use of sedative-hypnotics; subjects who have been taking a fixed dose of a sedative-hypnotic every day for a period of at least 30 days may be included provided that they continue the same regimen throughout the study.
7. Intermittent or chronic use of psychiatric medications (with the exception of antidepressants that have been stable for 3 months) or anti-epileptic drugs
8. Nursing home residents
9. Known allergy to oseltamivir phosphate or any of the inactive ingredients of Tamiflu®
10. Women who are pregnant, or planning to become pregnant, or who are lactating
11. Current alcohol or drug abuse or substance dependence
12. Participation in another clinical trial with an investigational drug within the last 30 days
13. Patients vaccinated for influenza within 6 months of study enrollment
14. In the Investigator's judgment, the subject will not be able to adhere to the protocol requirements or is not suitable for study participation for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. O'Mahony, M.D., Principal Investigator — London Road Diagnostic Clinic and Medical Centre
Locations (16):
- Canada (16):
  - Dr. Collette, Vancouver, British Columbia
  - Dr. Lai, Vancouver, British Columbia
  - Topsail Road Medical Clinic, St. John's, Newfoundland and Labrador
  - Moran Medical Centre, Collingwood, Ontario
  - Dr. Kanani, Etobicoke, Ontario
  - Dr. Herman, London, Ontario
  - Milestone Research, London, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - Family First Medical Centre, Orléans, Ontario
  - Steeple Hill Medical Centre, Pickering, Ontario
  - Dr. Martyn Chilvers - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Dr. Michael O'Mahony - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - DCTM Clinical Trials Group Ltd., Strathroy, Ontario
  - Dr. Gupta, Toronto, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Regina Medical Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oseltamivir | Standard of Care Alone
Started | 59 | 63
Completed | 59 | 62
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oseltamivir | Standard of Care Alone | Total
Number analyzed (Participants) | 59 | 63 | 122
Age, Continuous [Median (Full Range); unit: years] | 37.0 [17 to 66] | 32.0 [18 to 57] | 34.0 [17 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 43 | 49 | 92
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 59 | 63 | 122
Highest Education Level [Count of Participants; unit: Participants]
  Grade 5 - 11 | 7 | 3 | 10
  High School Graduate | 12 | 19 | 31
  1 - 3 Years College | 20 | 24 | 44
  Bachelor's Degree | 16 | 13 | 29
  Post-Graduate | 4 | 4 | 8
Current Smoker [Count of Participants; unit: Participants] | 7 | 14 | 21
Time from Symptom Onset [Median (Full Range); unit: hours] — Population: Data was not collected for 1 patient in each group in error
  hours
    number analyzed (Participants) | 58 | 62 | 120
    (all) | 33.8 [2.0 to 51.5] | 36.7 [5.3 to 55.0] | 35.0 [2.0 to 55.0]
Baseline Symptom Score [Median (Full Range); unit: symptom score] — Participants recorded the severity of 7 influenza symptoms (cough, nasal obstruction, sore throat, fatigue, headache, myalgia, and feverishness) using a 4-point scale (0, absent; 3, severe) each day for 14 days. Symptom severity was assessed by summing the severity rating (0-3) for the seven symptoms at each day.
  symptom score | 13 [3 to 21] | 14 [6 to 21] | 14 [3 to 21]
Body Temperature [Median (Full Range); unit: Degrees centigrade] | 38.1 [36.3 to 39.5] | 38.1 [36.5 to 39.3] | 38.1 [36.3 to 39.5]
Health Assessment Question [Median (Full Range); unit: Score] — Subjects rated their general health status each day using an 11-point VAS (0 = worst possible health; 10 = normal health for someone your age).
  Score | 3 [0 to 10] | 3 [0 to 10] | 3 [0 to 10]
Influenza Type [Count of Participants; unit: Participants] — Assessed through Rapid Antigen Test
  Participants
    Strain A | 53 | 52 | 105
    Strain B | 6 | 11 | 17
Cognitive/Mood Conditions [Count of Participants; unit: Participants]
  None | 53 | 60 | 113
  ADHD | 0 | 1 | 1
  Anxiety | 1 | 1 | 2
  Depression | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Attention Assessment
Description: Attention assessed using simple reaction time measured in milliseconds. Simple reaction time calculated as the mean of the following 2 sub-tests:
  * Reaction Time Subtest
  * Cued Reaction Time Subtest
  The lower the value, the better the attention.
Time Frame: Change from baseline at Day 4
Population: All randomised subjects for whom data was collected at both baseline and Day 4. Oseltamivir group: baseline data available for 58 of 59 randomised subjects and Day 4 data for 53 subjects (53 subjects analysed). Standard of Care Alone group: baseline data available for 61 of 63 subjects and Day 4 data for 55 subjects (55 subjects analysed).
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Oseltamivir | Standard of Care Alone
Number analyzed (Participants) | 53 | 55
milliseconds | -70.0 (10.9) | -39.7 (10.9)
Statistical Analysis 1: Comparison: Oseltamivir vs Standard of Care Alone; Test type: Superiority or Other; p = .0492, ANCOVA; LS Means Difference = -30.4, 95% CI 2-sided [-60.7 to -0.1] — The LS means for Standard of Care Alone was subtracted from that of Oseltamivir

2. Secondary Outcome: Change in Working Memory Assessment
Description: Working memory assessed with the Dot Memory Test.
  The higher the value, the better the working memory.
Time Frame: Change from baseline at Day 4
Population: All randomised subjects with data collected at both Baseline and Day 4. Oseltamivir Group: Baseline values collected for all randomized subjects (59); Day 4 data available for 54 subjects (54 analysed). Standard of Care Alone Group: Baseline values collected for all randomized subjects (63); Day 4 data available for 58 subjects (58 analysed)
Measure: Least Squares Mean (Standard Error); unit: Number of correct answers
Arm/Group | Oseltamivir | Standard of Care Alone
Number analyzed (Participants) | 54 | 58
Number of correct answers | 8.2 (0.95) | 4.4 (0.94)
Statistical Analysis 1: Comparison: Oseltamivir vs Standard of Care Alone; Test type: Superiority or Other; p = 0.0054, ANCOVA; LS Means Difference = 3.8, 95% CI 2-sided [1.14 to 6.42] — The LS means for Standard of Care Alone was subtracted from that of Oseltamivir

3. Secondary Outcome: Change in Processing Speed Assessment
Description: Processing speed assessed with the animal number decoding subtest
  The lower the value, the better the processing speed
Time Frame: Change from baseline at Day 4
Population: All randomized subjects for whom data was collected at both Baseline and Day 4. Oseltamivr Group: Baseline data available for all randomized subjects (59); Day 4 data available for 54 subjects (54 analysed). Standard of Care Alone Group: Baseline data available for all randomized subjects (63); Day 4 data available for 58 subjects (58 analysed).
Measure: Least Squares Mean (Standard Error); unit: Millliseconds
Arm/Group | Oseltamivir | Standard of Care Alone
Number analyzed (Participants) | 54 | 58
Millliseconds | -551.9 (77.6) | -555.8 (78.2)
Statistical Analysis 1: Comparison: Oseltamivir vs Standard of Care Alone; Test type: Superiority or Other; p = .9685, ANCOVA; LS Means Difference = 3.9, 95% CI 2-sided [-190.1 to 197.9] — The LS means for Standard of Care Alone was subtracted from that of Oseltamivir

4. Other Pre Specified Outcome: Change in Mood Assessment
Description: Mood was assessed using the Bond-Lader 10 cm (100 mm) visual analogue scales for mood (16 scales in total); factored for alertness (mean of 9 scales), calmness (mean of 2 scales) and contentment (mean of 5 scales).
  The range in score for each scale and for each factor (alertness, calmness and contentment) was 0 - 100 mm.
  Each scale was anchored such that the lower the value, the better the mood.
Time Frame: Change from baseline at Day 4
Population: All randomised subjects with data collected at both Baseline and Day 4. Baseline data was available for all randomized subjects in both groups; Day 4 data was available for 54 of 59 randomized subjects in the Oseltamivir Group (54 analysed) and for 58 of 63 randomized subjects in the Standard of Care Alone Group (58 analysed).
Measure: Least Squares Mean (Standard Error); unit: millimeter
Arm/Group | Oseltamivir | Standard of Care Alone
Number analyzed (Participants) | 54 | 58
millimeter
  Change in Alertness Assessment | 19.1 (1.4) | 17.2 (1.4)
  Change in Calmness Assessment | 3.0 (1.3) | 3.6 (1.2)
  Change in Contentedness Assessment | 16.3 (1.5) | 13.0 (1.5)
Statistical Analysis 1: Comparison: Oseltamivir vs Standard of Care Alone; Alertness: the higher the value, the greater the alertness; Test type: Superiority or Other; p = .3195, ANCOVA; LS Means Difference = 1.9, 95% CI 2-sided [-1.9 to 5.7] — The LS means for Standard of Care Alone was subtracted from that of Oseltamivir
Statistical Analysis 2: Comparison: Oseltamivir vs Standard of Care Alone; Calmness: the higher the value, the greater the calmness; Test type: Superiority or Other; p = .7219, ANCOVA; LS Means Difference = -.6, 95% CI 2-sided [-4.1 to 2.9] — The LS means for Standard of Care AL one was subtracted from that of Oseltamivir
Statistical Analysis 3: Comparison: Oseltamivir vs Standard of Care Alone; Contentedness: the higher the value, the greater the contentedness; Test type: Superiority or Other; p = .1162, ANCOVA; LS Means Difference = 3.3, 95% CI 2-sided [-.8 to 7.4] — The LS means of Standard of Care Alone was subtracted from that of Oseltamivir

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Oseltamivir | Standard of Care Alone
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/63
Other Adverse Events (participants affected / at risk) | 8/59 | 8/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir (N=59) | Standard of Care Alone (N=63)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor has not submitted a manuscript for publication for this multi-center study within 12 months of study completion/termination, the PI will be free to publish separately. Sponsor can review results communications prior to public release and can embargo communications for up to 90 days if the proposed publication contains information relating to patentable items. If Sponsor believes proposed communications contain any confidential information, Sponsor has the right to remove it.